CLINICAL TRIAL: NCT06814886
Title: Effects of Wearable Devices Initiates Behavioral Change Intervention on Body Composition, Physical Activity, Sleep Quality and Stress of Nurses in Hospital Working Place: A Randomized Controlled Trial
Brief Title: Effects of Wearable Devices Initiates Behavioral Change Intervention on Body Composition, Physical Activity, Sleep Quality and Stress of Nurses in Hospital Working Place
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, LO, YIPANG, Head Nurse in emergency department, SongShan Branch, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: A202405171
Record Dates: First submitted 2024-12-21; First posted 2025-02-07 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Nurse; Healthy Adult
Keywords: wearable device; behavioral change intervention; nurse; working place

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group(wearable devices to initiate behavioral intervention) (Experimental): 12 week wearable devices to initiate behavioral intervention including line APP recruited participants and give some behavior change advises, also give a APP-based motivational interviewing 15 minutes per week.
  Interventions: Behavioral: wearable devices to initiate behavioral intervention
- comparison group (wearable devices monitor only) (Active Comparator): 12 week wearable devices just monitor
  Interventions: Behavioral: 12 week wearable devices monitor

INTERVENTIONS:
Behavioral: wearable devices to initiate behavioral intervention — 12 week wearable devices to initiate behavioral intervention including line APP recruited participants and give some behavior change advises, also give a APP-based motivational interviewing 15 minutes per week.
  Arms: Intervention group(wearable devices to initiate behavioral intervention)
Behavioral: 12 week wearable devices monitor — 12 week wearable devices monitor physical activity and sleep quality only
  Arms: comparison group (wearable devices monitor only)

SUMMARY:
Background: Physically inactive and poor sleep quality are at increased risk for non-communicable diseases. Nurses were the most vulnerable inactive healthcare personnel who may not meet global physical activity recommendations because of complicated rotation shifts and heavy working loading. Wearable devices initiate behavior intervention combined with smartphone applications could offer new opportunities for social connection by a convenient way for nurses to improve physical activity and sleep quality.

Objectives: To evaluate the effects of wearable devices initiate behavioral intervention on body composition, physical activity, sleep quality and stress of nurses in hospital working place.

Method: This is a randomized controlled trial that will recruit 120 nurses and randomly assign them into two groups from a hospital working place. The nurses in the intervention group will receive 12-week wearable devices to initiate behavioral intervention. The nurses in the comparison group will only receive 12-week wearable devices monitoring. Data will be collected at baseline and 12-week and 24-week follow-up. The body composition will be measured by bioelectrical impedance analysis (BIA). The physical activity and sleep quality will be monitored by the Fitbit wearable device and application. The mediator parameter of the stress will be measured by salivary amylase activity (SAA). We will control the internal validity to assure the quality of training, treatment fidelity, identify barriers and facilitators of implementation, and assess participants' satisfaction. General estimating equations (GEE) will be applied to examine the effects of time and group interaction.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who give informed consent for this study and are 20 years old or older.
* Those who own a smartphone and are willing to join the study's LINE group.
* Individuals whose mobile application (APP) can synchronize with the Fitbit Charge 6 wearable device.
* Nurses who hold a nursing license and are working in a clinical setting.

Exclusion Criteria:

* Individuals unable to provide informed consent for this study and are younger than 20 years old.
* Those who do not own a smartphone.
* Individuals who do not have a nursing license or are not employed in a clinical setting as a nurse.
* Participants who are already involved in other health promotion or exercise training studies.
* Nurses who are currently pregnant.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Physical activity (subjective) | From enrollment to the end of treatment at 12 weeks, and 24 weeks follow up
  Measurement Tool: International Physical Activity Questionnaire short form - Taiwan version
Physical activity (objective) | From enrollment to the end of treatment at 12 weeks, and 24 weeks follow up
  Measurement Tool: Wearing Fitbit Charge 6 HR to collect physical activity and sleep quality related data.

SECONDARY OUTCOMES:
Sleep quality (objective) | From enrollment to the end of treatment at 12 weeks, and 24 weeks follow up
  Measurement Tool: Wearing Fitbit Charge 6 HR to collect physical activity and sleep quality related data.
sleep quality (subjective) | From enrollment to the end of treatment at 12 weeks, and 24 weeks follow up
  Measurement Tool:Chinese version of the Pittsburgh Sleep Quality Index (CPSQI)
Body composition | From enrollment to the end of treatment at 12 weeks, and 24 weeks follow up
  Measurement Tool: Inbody 270 Body Composition Analyzer
Stress | From enrollment to the end of treatment at 12 weeks, and 24 weeks follow up
  Measurement Tool: Nipro Salivary Amylase Activity Monitor and enzyme-linked immunosorbent assay (ELISA) will be utilized to quantify the levels of irisin, IL-6, and BDNF in serum samples, allowing for the assessment of immune stress values.

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Background: Physically inactive and poor sleep quality are at increased risk for non-communicable diseases. Nurses were the most vulnerable inactive healthcare personnel who may not meet global physical activity recommendations because of complicated rotation shifts and heavy working loading. Wearable devices initiate behavior intervention combined with smartphone applications could offer new opportunities for social connection by a convenient way for nurses to improve physical activity and sleep quality.
  Objectives: To evaluate the effects of wearable devices initiate behavioral intervention on body composition, physical activity, sleep quality and stress of nurses in hospital working place.
  Method: This is a randomized controlled trial that will recruit 120 nurses and randomly assign them into two groups from a hospital working place. The nurses in the intervention group will receive 12-week wearable devices to initiate behavioral intervention. The nurses in the comparison group will
Supporting Information: Study Protocol
Time Frame: 2025/3/1 will be available and end in 2027/3/1